CLINICAL TRIAL: NCT05925777
Title: Plantar Fasciitis Treatment: Influence of the Possible Presence of Subchondral Bone Edema
Acronym: THEAL-F
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: THEAL-fasc
Record Dates: First submitted 2023-06-13; First posted 2023-06-29 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Fasciitis, Plantar
Keywords: laser; foot; ankle; pain
MeSH Terms: conditions — Fasciitis, Plantar; Pain | interventions — Lasers

STUDY DESIGN:
Intervention Model Description: randomized prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- experimental group (Experimental): The protocol provides for the administration of 10 polymodal high energy laser therapy sessions, to be carried out every other day. The THEAL device (Mectronic, Bergamo) allows to deliver 4 wavelengths (650 nm, 810 nm, 980 nm and 1064 nm), with continuous and pulsed mode, with power up to 20 W.
  Patients will perform stretching exercise like those of the control group.
  Interventions: Device: THEAL (Mectronic, Bergamo)
- Control group (No Intervention): Patients will perform four daily stretching exercises (three sets of 30 seconds), for 6 weeks.
  1. Hamstring and ankle plantar flexor stretch (straight leg raise in supine position)
  2. self-stretching of the surae muscles: the patient bends forward in a standing position with the affected foot farthest from the wall, keeping the heel on the floor; 3. the soleus muscle is exercised with the knee flexed and the gastrocnemius muscle with the knee extended
  4. Plantar fascia self-stretch: In a seated position, the patient crosses the affected foot over the contralateral thigh and passively extends the metatarsophalangeal joints .
  In the first session, the volunteers will be trained on how to perform the exercises correctly and will be monitored once a week.

INTERVENTIONS:
Device: THEAL (Mectronic, Bergamo) — laser therapy high intensity
  Other Names: laser
  Arms: experimental group

SUMMARY:
Standard treatments of plantar fasciitis include stretching exercises of the posterior muscle chain and plantar fascia, taking anti-inflammatories, cortisone infiltration or biostimulation with physical therapies (low energy laser therapy, shock waves, ultrasound therapy, etc.). In non-responsive forms to conservative treatments, surgical treatment can be undertaken.

Laser therapy is indicated for plantar fasciitis, in particular for its biological anti-inflammatory, anti-edema and reparative effects on the plantar fascia; to date, the potential effects also on the underlying bone edema component, when present, which aggravates and self-maintains the ongoing pathology are not known.

DETAILED DESCRIPTION:
Plantar fasciitis is one of the most common causes of heel pain; the pain is more intense in the morning, tends to decrease during the day with movement, to flare up after sitting for a long time. It presents itself as inflammation and contextual degeneration of the insertion of the fascia that covers the muscles present at the level of the sole of the foot, with progressive evolution and possible calcification of the insertion. The incidence is between 9 and 20% of the population, with a higher incidence in middle-aged obese women and in young male runners. The diagnosis makes use of radiography, to verify any local deformities or the presence of the subcalcaneal spur, and ultrasound, to investigate the integrity of the fascia and its thickening. MRI images are useful for better studying the heel bone and plantar fascia, especially for discerning other various causes of heel pain, including stress fractures, tarsal tunnel syndrome, and Achilles tendinopathy. Signal changes with bone edema are sometimes found in association with plantar fasciitis and may be indicative of or represent the result of avulsive trauma, stress, intraspongious fractures or a combination of these situations. These MRI images are similar to those described in the elbow in some patients with epicondylitis, where overuse can cause increased bone edema on T2-weights. Previous studies have shown the presence of bone edema at the level of the heel on MRI in 35% of patients with plantar fasciitis. Plantar fascia evaluation with a dedicated magnetic resonance scanner in weight-bearing position: our experience in patients with plantar fasciitis and in healthy volunteers. Maier et al demonstrated that the presence of calcaneal bone edema is a highly predictive factor for improved response to shock wave treatment. Often the finding of a thickening of the fascia and the signal changes of the soft tissues do not correlate with the clinical response, while the presence of bone edema is highly predictive (positive predictive value 0.94, sensitivity 0.89, specificity 0.8).

ELIGIBILITY:
Inclusion Criteria:

1. history of heel pain for at least 3 months prior to enrollment,
2. Pain on palpation of the medial calcaneal tubercle or proximal plantar fascia,
3. plantar fascia thickness of 4.0 mm or greater.

Exclusion Criteria:

1. age below 18 years of age
2. history of systemic disease
3. pregnancy
4. Previous surgery on the lower limbs
5. diagnosis of fibromyalgia, neurological disease, Achilles tendinopathy, metatarsalgia, acute ankle sprain, tarsal tunnel syndrome, or heel joint syndrome
6. body mass index (BMI) greater than 35 kg/m2
7. wounds, infections in the treatment area
8. altered sensation in the treatment area
9. skin pigmentation alterations in the area to be treated (tattoo, dyschromia)
10. metal implants in the treatment area
11. History of oral or injected corticosteroid therapy within the past six weeks
12. Diagnosis of neurological heel pain (radiculopathy)
13. diagnosis of systemic inflammatory arthritis (rheumatoid arthritis, etc.)
14. other acute pathologies (febrile fever, cold, etc.) requiring treatment
15. other painful conditions requiring painkillers (toothache, back pain, etc.)
16. neoplasms
17. cardiac pacemaker or other device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
recovery of pain | change between baseline to 2 months
  The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain."
recovery of pain | change between baseline to 6 months
  The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain."

SECONDARY OUTCOMES:
functional recovery | change between baseline to 2 months
  The Foot Function Index (FFI) measures the effect of foot problems on function in terms of pain and disability.The scores range from 0 to 100; the higher the score, the more limitation/pain/disability is present. The scores range from 0 to 100; the higher the score, the more limitation/pain/disability is present.
functional recovery | change between baseline to 6 months
  The Foot Function Index (FFI) measures the effect of foot problems on function in terms of pain and disability.The scores range from 0 to 100; the higher the score, the more limitation/pain/disability is present. The scores range from 0 to 100; the higher the score, the more limitation/pain/disability is present.
perception of clinical improvement | change between baseline to 2 months
  Maudsley and Roles scale scores range from 0-4 points for excellent to poor
perception of clinical improvement | change between baseline to 6 months
  Maudsley and Roles scale scores range from 0-4 points for excellent to poor

OTHER OUTCOMES:
band thickness | change between baseline to 2 months
  ultrasound image to measure of fascia thickness, measured in mm
band thickness | change between baseline to 6 months
  ultrasound image to measure of fascia thickness, measured in mm
presence of edema | change between baseline to 2 months
  MRI image to verify the presence or absence of bone edema (dichotomous answer)
presence of edema | change between baseline to 6 months
  MRI image to verify the presence of absence or bone edema (dichotomous answer)

CONTACTS AND LOCATIONS:
Locations (1):
- Angela Notarnicola, Bari, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] DiGiovanni BF, Nawoczenski DA, Lintal ME, Moore EA, Murray JC, Wilding GE, Baumhauer JF. Tissue-specific plantar fascia-stretching exercise enhances outcomes in patients with chronic heel pain. A prospective, randomized study. J Bone Joint Surg Am. 2003 Jul;85(7):1270-7. doi: 10.2106/00004623-200307000-00013. PMID 12851352